CLINICAL TRIAL: NCT06680752
Title: A Phase 1/2, Open-label, Multicenter Trial to Assess the Safety and Efficacy of ARD103 in Patients With Relapsed or Refractory Acute Myeloid Leukemia or Myelodysplastic Syndrome
Brief Title: Clinical Study of ARD103 CAR-T Therapy for Patients With R/R AML or MDS
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARCE Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD103_ARCE-CL-P-001
Record Dates: First submitted 2024-10-29; First posted 2024-11-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia, in Relapse; Acute Myeloid Leukemia Refractory; MDS (Myelodysplastic Syndrome)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- phase 1 (Dose Escalation) and phase 2 (Dose Expansion) (Experimental): In Phase 1, three escalating dose levels will be tested using the 3 + 3 design. The MTD and RP2D will be identified.
  The Phase 2 will be conducted in 2 stages. In Stage I, evaluable participants from Phase 1 treated at RP2D will be enrolled. And the enrollment will continue into Stage II (additional evaluable participants) at the maximum RP2D participants for preliminary overall assessment of efficacy and safety.
  Interventions: Biological: ARD103; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: ARD103 — ARD103 autologous CAR-T cell therapy targeting CLL-1, single iv. infusion
Drug: Cyclophosphamide — iv administration for lymphodepletion
Drug: Fludarabine — iv administration for lymphodepletion

SUMMARY:
This is a phase I/2, interventional, open-label, multicenter study to assess the safety and efficacy of ARD103 in patients with relapsed or refractory acute myeloid leukemia or myelodysplastic syndrome.

DETAILED DESCRIPTION:
The investigational product (IP) for this study is ARD103, a C-type lectin-like molecule-1 (CLL-1) autologous chimeric antigen receptor T-cells (CAR-T). CLL-1 is highly expressed on both myeloid blasts and leukemia stem cells (LSCs) but is absent on normal hematopoietic stem cells (HSCs), suggesting CLL-1 as an excellent therapeutic target for AML and hence other potential myeloid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of AML with either refractory or relapsed disease or diagnosis of MDS and ≥ 5% BM blasts
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic status:

  * Absolute lymphocyte count (ALC) > 100/mm3
* Adequate renal, hepatic, cardiac and pulmonary function:

  * ALT and AST < 3.0 × the ULN
  * Creatinine clearance ≥ 45.0 mL/min as estimated by Cockcroft-Gault and independent dialysis
  * Total bilirubin ≤ 2.0 mg/dL
* Pregnancy testing: females of childbearing potential must have a negative serum or urine pregnancy test
* Contraception: males and females of childbearing potential must agree to use an effective method of contraception
* Participant is capable of giving signed informed consent

Exclusion Criteria:

* Participants with acute promyelocytic leukemia
* Presence of active and clinically relevant central nervous system (CNS) disorder
* Autoimmune disease requiring immunosuppressive treatment
* Participants with known hepatic bridging cirrhosis
* Currently active infection with hepatitis B or C
* Previous treatment with investigational gene or cell therapy (including CAR therapy)
* Any active acute GvHD or systemic treatment of more than 10 mg prednisone daily (or equivalent)
* Previous chemotherapy including biologic/targeted therapy or immunological agents directed to the pathology within 14 days prior to screening and all along the study duration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 days post ARD103 infusion
  The records of AEs and severity following the first infusion of ARD103.
To determine the RP2D of ARD103 | 28 days post ARD103 infusion
  RP2D of ARD103 following a 3+3 dose escalation schema (Phase 1)
To evaluate overall response rate (ORR) | Up to 24 months
  The ORR will be evaluated by European Leukemia Net (ELN) criteria

SECONDARY OUTCOMES:
Overall Survival (OS) | First infusion date of ARD103 up to 15 years
  OS is defined as the time from ARD103 infusion to the date of death from any cause.
Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from the infusion of ARD103 infusion to the first recorded response of disease progression, relapse, or death due to any cause, whichever occurs first.
Time to best response | First infusion date of ARD103 up to 24 months
  Time to best response is defined as the time from the infusion of ARD103 to the BOR.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Novant Health Cancer Institute, Charlotte, North Carolina
  - Novant Health Cancer Institute, Winston-Salem, North Carolina
  - MD Anderson Cancer Center, Houston, Texas